CLINICAL TRIAL: NCT04966468
Title: Look of Life 2.0. Virtual Reality for Cancer Patients in Home Palliative Care
Acronym: LOL2020_ANT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione ANT Italia ONLUS (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Principal Investigator, Vittoria Sichi, Psychologist, Psychoterapist, Fondazione ANT Italia ONLUS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 542-2019-OSS-AUSLBO
Record Dates: First submitted 2021-06-01; First posted 2021-07-19 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Oncological Patients; Virtual Reality
Keywords: Anxiety; Cancer; Depression; Digital health care; Immersive technology; Pain; Palliative care; Virtual reality
MeSH Terms: conditions — Anxiety Disorders; Neoplasms; Depression; Pain

STUDY DESIGN:
Intervention Model Description: The proposed investigation is a randomized, controlled, non-profit, single-center exploratory interventional study without drugs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Group (Experimental): Patients will be given the VR headset with non-interactive and interactive contents at home for four days
  Interventions: Device: Virtual Reality
- CTR group (Active Comparator): Patients will be given a tablet at home for four days with relaxing non-interactive 2D videos with natural and artistic scenarios
  Interventions: Other: Control

INTERVENTIONS:
Device: Virtual Reality — The Lenovo Mirage Solo Headset will be kept at home by the patient for the duration of the study (4 days). The VR headset will be equipped with 10 non-interactive videos and a short interactive game. The videos and the game are characterized by relaxing scenarios. The game will require the active interaction of the patient. At the end of the observational period, the investigator will download the usage data to detect information about the patient's use. Before and after each use of the VR headset, the patient will be asked to fulfil the Edmonton Symptom Assessment Scale (ESAS). On T0, the patient will be asked to wear a wearable device, the Empatica E4 wristband measuring physiological parameters. On day T1, the patient will return the VR headset and the wristband to the investigator and will fulfil again the HADS and BPI questionnaires.
  Arms: VR Group
Other: Control — The investigator will illustrate to the patient how to use the tablet for watching videos, suggesting using it especially in moments of psycho-physical discomfort. The tablet will be given to the patient for the duration of the study (four days). The tablet will be equipped with 10 non-interactive 2D videos characterized by relaxing settings with natural or artistic scenarios, giving a "passive" use to the patient. Before and after each use of the tablet, patient has to fullfil the ESAS digitally inserted into the tablet. Patient can answer by selecting the answer on the touchscreen. Without filling the scale, the patient will not be able to access the videos inserted in the tablet. On day T1, patient will return the tablet to the investigator and fill out the HADS and BPI questionnaires.
  Arms: CTR group

SUMMARY:
Oncological disease, in addition to undermining the physical health and autonomy of the patient, is often accompanied by significant anxious and depressive symptoms that can compromise the quality of life of both patient and his/her family, hindering the adherence to treatment, the effectiveness of therapies and worsening the clinical prognosis.

Several studies confirm that a large number of cancer patients experience severe levels of psychological distress, with an average prevalence of any mood disorder ranging from 29% in palliative care to 38% in oncological and hematological settings.

The advanced stages of the disease are characterized by a progressive loss of functional autonomy, forcing the patient to a condition of isolation and both sensory and relational deprivation. The reduction of the occasions in which it is possible to experience positive emotions and meaningful social interactions often corresponds to an intensification of obsessive worries and thoughts, which in turn increase stress and connect to further negative emotional experiences. Thus the patient can be trapped in a vicious circle, that might increase the worsening of quality of life.

In the last years, alongside traditional interventions, the effectiveness of interventions based on the use of immersive audiovisual technologies has been tested, such as the use of virtual reality (VR), which have the ability to emotionally involve the person, capture his/her attention and direct it towards positive stimuli, without particular effort to be used.

Compared to 2D or 3D videos, VR gives to the user a "greater degree of presence", giving the impression of being immersed in a reality different from the real one. Unlike any other form of psychological intervention, VR does not require special training to be used and has the advantage of being used even in situations of poor mobility or attention capacity.

Available literature shows how the use of VR for cancer patients is a widespread practice that can be considered an additional psychological technique. Several studies showed that VR can help in decreasing the psychophysical symptoms usually experienced by cancer patients in different settings (e.g., chemotherapy sessions, invasive medical procedures, and hospitalization). However, up to now, there are no studies in the scientific literature on the use of VR in the context of home palliative care. In this setting, it could be extremely interesting to test the effectiveness of this innovative technology, due to its growing diffusion and accessibility.

The present study is aimed at assessing the effects of VR in cancer patients followed by ANT Foundation home palliative care program. The VR headset will be kept at the patients' home so that he/she can use it in moments of greatest psychophysical discomfort (e.g., pain peaks, moments of anxiety or sadness). The VR will contain both non-interactive and interactive contents, the last ones specifically developed for ANT patients.

DETAILED DESCRIPTION:
Background Many cancer patients experience severe levels of psychological distress, with a percentage varying from 10-15% to 20-40% (Mitchell et al., 2011; Shim et al., 2018). The average prevalence of mood disorders ranges from 29% in palliative care settings to 38% in cancer and hematological contexts (Jacobsen et al., 2005). In addition to the emotional distress, the advanced stages of the disease often imply a progressive loss of functional autonomy (Dong et al., 2016). This put the patient in a status of deprivation and forced isolation from relational and social aspects that were hitherto in their lives. This psychological distress naturally adds to the burden of the physical symptoms caused by the disease and/or invasive therapies, above all pain.

In the last years, technological innovation has allowed new solutions to meet old and emerging needs in the healthcare field. One of these is represented by Virtual Reality (VR), a non-invasive simulation technology that allows the user to be immersed in a multisensory experience. VR technologies can emotionally involve the patients, inducing a positive mood and allowing them to feel like a part of the virtual environment (Malloy and Milling, 2010; Pourmand et al., 2018; Ahmadpour et al., 2019). The distraction effect is recognized to be the primary principle underlying the effectiveness of VR (Schneider et al., 2004; Malloy and Milling, 2010; Wiederhold et al., 2014; Bani Mohammad and Ahmad, 2019), as it is capable of diverting patient's attention from his or her current clinical condition. Natural contents have been shown to induce relaxation and restore work productivity, based on the Attention Restoration Theory (Kaplan, 1995; Berto, 2005; Anderson et al., 2017). Moreover, water scenes with views and sound seem to be more appreciated than scenes without water (White et al., 2010; Anderson et al., 2017). Additionally, interactive contents could be even more effective in their distraction-based effect than contents that only require passive observation (Wiederhold and Wiederhold, 2007; Shahrbanian et al., 2012; Wender et al., 2019). VR-based interventions are a convenient solution, as they do not require complicated training to be used and can be employed in case of low mobility conditions.

VR has been used as an adjuvant treatment in various clinical conditions to relieve pain, anxiety, and depression (Dascal et al., 2017; Fodor et al., 2018), during invasive procedures (Hoffman et al., 2011; Shetty et al., 2019; Brown and Foronda, 2020), for chronic pain management (Wiederhold et al., 2014; Pekyavas and Ergun, 2017) and in rehabilitation settings (Shahrbanian et al., 2012; Lee et al., 2015). It has been extensively employed in promoting cancer patients' psychological well-being (Chirico et al., 2016; Zeng et al., 2019; Ioannou et al., 2020). Previous studies assessed the effects of VR in relieving cancer-related symptomatology mainly in clinical settings (Li et al., 2011; Baños et al., 2013; Mosadeghi et al., 2016; Bani Mohammad and Ahmad, 2019), alleviating anxiety and improving mood states. Studies in palliative care (PC) have proven the acceptability of VR interventions (Oyama, 1997; Brungardt et al., 2020; Weingarten et al., 2020) and their effect in reducing short-term symptoms (i.e., pain, drowsiness, lack of appetite, shortness of breath, depression, anxiety, and well-being) (Niki et al., 2019; Johnson et al., 2020).

The evidence about the use of VR in a home PC program is still insufficient. To fill this gap, the National Tumor Assistance Foundation (ANT), a non-profit organization working in Italy in the field of home PC and pain management, conducted a pilot study to test the feasibility of VR interventions for cancer patients assisted at home (Varani et al., 2018). This was the first attempt to introduce VR interventions in home-PC settings, obtaining promising results: most participants (73%) declared that they would be willing to keep a VR headset at home; patients showed a 20% decrease in anxiety and depression and a significant reduction of perceived pain and fatigue symptoms. As a further outcome, ANT collected patients' preferences as the output of a focus group and semi-structured interviews: all patients declared to prefer natural and relaxing scenarios, 36% expressed a preference for interactive videos, while 33% wanted to see videos as simple observers (Sichi et al., 2019).

After these encouraging results, ANT introduced the VR headset with interactive and non-interactive contents in its home-care practice.

VR use is not intended as a substitute for psychological support, but as an additional and complementary intervention to allow the patient to have moments of leisure and distraction from their psycho-physical condition.

Study design The proposed investigation is a randomized, controlled, non-profit, single-center exploratory intervention study without drugs.

The study is aimed to evaluate the effect of immersive VR use on the psycho-physical symptoms of cancer patients assisted by the ANT Foundation home palliative care program.

Patients who meet the inclusion criteria will be randomly assigned to one of the following two groups:

Experimental group (VR group): patients will be given the VR headset with non-interactive and interactive contents at home for four days

Control group (CTR group): patients will be given a tablet at home for four days with relaxing non-interactive 2D videos with natural and artistic scenarios.

VR and CTR patients will undergo the same tests in the same time frame.

Primary outcome

- Anxiety and depression levels.

Secondary outcome

* Pain.
* Short-term psychophysical symptoms.
* To identify the type of immersive VR content and the average VR time-usage resulting most beneficial for the home palliative care cancer patient.

Study population and setting The study population consists of cancer patients assisted by the home palliative care program of the ANT Foundation in Bologna city and surrounding areas (Italy). The study will take place directly at the patients' homes.

Randomization The investigators (ANT psychologists), after having exposed the study, will ask the ANT physicians to identify patients who meet eligibility criteria among their assisted ones. The physicians will explain the study to eligible patients and, if they show interest to participate, they will be contacted by the psychologist. Patients will be randomly assigned by the Research Department of the ANT Foundation to the VR group (30 patients) or the CTR group (30 patients) by randomization using a series of random numbers generated by Excel. Investigators that will run the statistical analysis will be blinded to the randomization procedure.

Procedure and measures The study will last for four days for each patient. On the first day (T0) each subject will be fully explained the study, given the specific information, and asked to sign the informed consent. The psychologist, after filling the socio-demographic and clinical data sheet, will ask the participant to answer the following set of validated questionnaires which will then be administered for the second time at the end of the 4 days of observation (T1). The procedure takes approximately 30 minutes at T0, and 10 minutes at T1.

Hospital Anxiety and Depression Scale (HADS)

Brief Pain Inventory (BPI)

VR Group. After having filled the questionnaires, the investigator will show the patient how to use the VR headset, suggesting using it especially in moments of psycho-physical discomfort. In this study, a Lenovo Mirage Solo Headset, together with the wireless Daydream motion controller, will be used. The VR headset will be kept at home by the patient for the duration of the study (i.e., four days). The VR headset will be equipped with 10 non-interactive videos and a short interactive game. The videos are characterized by relaxing scenarios (e.g., beach, sunset over the sea), giving a "passive" use to the patient. The game is also characterized by a relaxing scenario and it will require the active interaction of the patient. At the end of the observational period, the investigator will be able to download the usage data to detect useful information, i.e., knowing if the patient has used the VR headset to view interactive or non-interactive contents and the time of use. Before and after each use of the VR headset, the patient will be asked to fulfill the Edmontom Symptom Assessment Scale (ESAS), an internationally validated rating scale used to assess the impact of the main symptoms on the quality of life in patients in palliative care. The ESAS is composed of some numerical rating scales (NRS) relating to specific symptoms ranging from 0 (absence of the symptom) to 10 (worst symptom severity). The evaluated symptoms are pain, nausea, depression, anxiety, drowsiness, lack of appetite, malaise, and shortness of breath. In order to ensure the correct completion of the ESAS scales, it will be digitally inserted directly into the VR headset, and the patient can answer by selecting the answer navigating with the controller. Without filling the scale, the patient will not be able to access the contents. On T0, the patient will be also asked to wear, for the entire duration of the study, a wearable device, the Empatica E4 wristband, that measures several physiological parameters (skin conductance, heart rate, skin temperature) associated with painful experiences and anxious symptoms. Patients will be also provided with a short paper diary in which they can record any pain or anxiety peak experienced during the day, as well as any drug taken to overcome such moments of psychophysical discomfort (e.g., painkillers, benzodiazepines). On the second day, the investigator goes back to the patient in order to download data from Empatica E4 wristband and recharge it. On day T1, the patient will return the VR headset and the wristband to the investigator and will complete again the HADS and BPI questionnaires.

CTR group. After having administered the questionnaires, the investigator will illustrate to the patient how to use the tablet for watching videos, suggesting using it especially in moments of psycho-physical discomfort. The tablet will be given to the patient for the duration of the study (four days). The tablet will be equipped with 10 non-interactive 2D videos characterized by relaxing settings with natural or artistic scenarios, giving a "passive" use to the patient. Before and after each use of the tablet, the patient has to complete the ESAS digitally inserted into the tablet. The patient can answer by selecting the answer on the touchscreen. Without filling the scale, the patient will not be able to access the videos inserted in the tablet. On day 4 (T1), the patient will return the tablet to the investigator and fill out the HADS and BPI questionnaires.

Security precautions The risk analysis, and the subsequent control measures, are based on the device documentation provided by the manufacturer, the scientific literature, and the evidence and experience gained with the Look of Life pilot study, conducted by ANT and the University of Padova. In order to cover potential risks for patients, ANT Foundation has taken out a study-specific insurance policy.

* Risk from electromagnetic emissions from VR headset. The investigators consider this risk to be an acceptable level, given the European Certification (EC) of the device. The device complies with the European Directive 2014/53/EU. Its Specific Absorbance Rate (SAR) is 0.097 W/Kg (maximum for European standards for mobile devices 2 W/Kg).
* Mechanical risk. When wearing the device, the user is not able to see the real surrounding space and could therefore trip or bump into objects. The instructions suggest using the headset in an environment free from obstructions such as objects and furniture. The device also gradually begins to obscure the view when the user moves more than 0.4 m from the position selected as the central position and darkens completely beyond 0.8 m. As an additional safety measure, investigators will instruct participants to use the headset only when seated, thereby reducing the risk to an acceptable level.
* Nausea and motion sickness. In some cases, especially with particular contents and in predisposed subjects, VR can elicit some episodes of nausea reported in the scientific literature. However, in the pilot study conducted by ANT and the University of Padova, no patient reported side effects due to the use of the VR headset. The investigator will immediately stop the study if the patient shows any episodes of nausea or motion sickness. The videos have been selected as they contain minimal stimuli that can elicit motion sickness or emotional distress. All videos and interactive content within the VR headset were created by Immerxive, a company specialized in the creation of multimedia content, under the supervision of the ANT psychologists who had participated in the pilot study. Furthermore, suffering from nausea or motion sickness are also exclusion criteria for participation in the study.
* Risk of infection. The VR headset is worn in contact with the user's face, therefore it could be a vehicle for infective agents among the study participants. Cleaning procedure will adhere to the guidelines of the regional health and social agency of Emilia Romagna (Agenzia sanitaria e sociale regionale dell'Emilia Romagna) concerning the disinfection of medical devices and equipment. The investigators considered the headset, as it is in contact with the user's face, as an oxygen therapy mask, for which the disinfection with chlorine derivatives at a concentration of 0.1% is recommended. Before each use from each subject, the VR headset will be disinfected with disposable sanitary wipes and the lenses will be cleaned with specific alcohol-based products. The controller, the tablet for the control group, and the wristband will be also disinfected after each patient use.
* Seizures. Diagnosis of epilepsy, other neurological diseases, and sensitivity to flashing lights are exclusion criteria for participation in the study.
* Eye fatigue, skin problems. ANT investigators, as already present in the device user manual, advise participants against prolonged use and indicate to wear the headset on clean and dry skin, and stop using it in case of signs of irritation, swelling, eczema, or itching.
* Fraudulent access to data. The headset and the tablet record information on the time of use of the device and on the assessments on the clinical scales carried out before and after each session. As a control measure, the data are stored on the device anonymously. Once the experimental phase for each subject is completed, the investigator sends a .txt file to the email address specifically set up for receiving these reports from the device restricted area (accessible only for the investigators by providing a password). Once archived, the file within the device is deleted before the next use by a new participant in the study.

For both groups, patients are aware through informed consent about the possible adverse events (i.e., nausea, dizziness, motion sickness). The investigator keeps in contact with patients for the whole study duration to immediately record any adverse event.

To cover the risks of adverse events described below, ANT Foundation has subscribed a study-specific insurance policy.

Sample size The sample size was evaluated using G*power software with a-priori power analysis for a one-sample Mann-Whitney-Wilcoxon test. Considering an α = 0.05 and a power 1-β = 0.80 with an effect size of 0.80, two groups of 27 patients each need to be enrolled for the study. Considering a 10% dropout rate, the study aims to recruit a total of 60 patients (30 patients for the VR group + 30 patients for the CTR group).

Statistical analysis Statistical analysis will be conducted on the data after their anonymization. An investigator is in charge of anonymization and blinding to groups patients allocation. The anonymized and blinded data will be passed to the investigators in charge of data analysis. Anonymized data will be stored within the Research Department of ANT Foundation in an ad-hoc safe electronic database.

A descriptive analysis of the socio-demographic and clinical data of the patients at T0 will be considered: age, marital status, educational qualification, occupation, neoplasm primary site, the extent of the neoplasm, Karnofsky index, and drugs intake. Comparison analysis on changes in anxiety, depression, and pain will be performed using mixed-effects models or non-parametric statistical tests (e.g., Mann-Whitney-Wilcoxon). Similarly, changes in short-term psychophysical symptomatology before and after the use of the VR headset/tablet will be evaluated using mixed-effects models. The sociodemographic and clinical characteristics of the subject, the type of VR content, and the usage times will be carried out by adding covariates to the mixed-effects models. The analysis will follow the "intention to treat" analysis.

Timeline

The project is scheduled in 3 phases:

* Phase 1 (1 month) - Training and patients selection - After the registration of the study protocol, the investigators (ANT psychologists) will explain to the ANT physicians the rationale, the protocol, the eligibility criteria of the study and will verify with each of them the presence of patients that can be enrolled.
* Phase 2 (8 months) - Recruitment and data collection - Each physician will contact eligible patients and ask them to participate. If the patient agrees, the physician will provide the patient contact data to the psychologist who will contact him/her. The psychologist will bring the VR headset or the tablet to the patient's home and will enroll the patient in the study.
* Phase 3 (4 months) - Statistical analysis and publication - The data collected will be statistically processed by the Research Department of the ANT Foundation for publication in scientific journals of the sector. The publication of the trial results will follow the CONSORT checklist.

Data management

* Data from electronic clinical scale assessment. Patients from both groups are asked to fulfill the Edmonton Symptoms Assessment Scale before and after each use of the device. These data are stored locally in the device and then sent to a pre-specified email address specifically generated for this purpose. ANT investigator can access the data within the device by entering the restricted area with a password.
* Data from Empatica E4 wristband. Physiological signals recorded by the smart wristband are recorded and stored locally. On day 2 and day 4, the investigator download data to the Empatica proprietary cloud platform and then locally
* Electronic records. Fulfilled questionnaires at T0 (day 1) and T1 (day 4) (HADS and BPI) and information about information by the Case Report Form (CRF) are reported digitally in a folder shared with all the investigators. Data are completely anonymized.

ELIGIBILITY:
Inclusion Criteria:

* able to understand the objectives of the study and to sign the informed consent;
* patient in ANT assistance, and not excluded according to the exclusion criteria listed below;
* age 18-70 years;
* able to speak and understand the Italian language.

Exclusion Criteria:

* cognitive disorders;
* epilepsy, dementia or other neurological disorder that could prevent the use of a VR technology;
* severe visual impairment;
* sensitivity to flashing lights;
* recent heart attack (less than 1 year);
* fixed breathing device;
* eyes or faces injuries preventing the correct use of virtual reality headset;
* unable to understand and speak the Italian language;
* unable to perform movements with the head or body to follow the 360 ° video;
* nausea or motion sickness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of anxiety and depression levels. | Day 1 and day 4
  This outcome will be measured by evaluating the scores obtained by Hospital Anxiety and Depression Scale (HADS) at day 1 (T0) and day 4 (T1). Two separate scores will be evaluated, one for anxiety and the other for depression, ranging from a minimum of 0 to a maximum of 21 points

SECONDARY OUTCOMES:
Change of pain experienced in the 24 hours prior to day 1 (T0) and and day 4 (T1). | Day 1 and day 4
  The measured outcome will be the score reported using the Brief Pain Inventory (BPI) questionnaire from a minimum of 0 to a maximum of 10 with respect to the worst, mildest, and average pain in the 24 hours preceding the administration of the questionnaire and the current one referred to when it was filled out.
Change of short-term psychophysical symptoms immediately after using the VR headset/tablet. | Day 1, day 2, day 3 and day 4.
  This reduction will be measured by comparing the scores before and after each use of the VR headset/tablet for each Edmonton Symptom Assessment System (ESAS) item. ESAS questionnaire is used to rate the intensity of nine common symptoms experienced by cancer patients (pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being and shortness of breath). Patients can rate the severity at the time of assessment of each symptom from 0 to 10 on a numerical scale, 0 meaning that the symptom is absent and 10 that it is of the worst possible severity.
To understand which type of immersive VR content is most beneficial for the home palliative care cancer patient | Day 1, day 2, day 3 and day 4.
  This outcome will be evaluated by comparing the results obtained on the ESAS scale before and after the use of non-interactive and interactive contents.
To understand the average usage of the VR headset that are the most effective. | Day 1 and day 4
  Usage times will be evaluated in association with the variation of the HADS score from day 1 (T0) to day 4 (T1).

CONTACTS AND LOCATIONS:
Overall Officials: Vittoria Sichi, Principal Investigator — Fondazione ANT Italia ONLUS
Locations (1):
- Fondazione ANT Italia ONLUS, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No